CLINICAL TRIAL: NCT01628133
Title: Packed Red Blood Cell Transfusion and Intestinal Blood Flow in Preterm Infants
Brief Title: Packed Red Blood Cell Transfusion and Intestinal Blood Flow in Preterm Neonates
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Aaron Pitzele, MD, Associte Professor of Pediatrics, St. Louis University
Other Study IDs: '20969
Record Dates: First submitted 2012-06-01; First posted 2012-06-26 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Intestinal Blood Flow
Keywords: Transfusion; Neonate; Infant, Very Low Birth Weight; Patent Ductus Arteriosus; Packed Red Blood Cell
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- blood transfusion group
  Interventions: Procedure: ultrasound

INTERVENTIONS:
Procedure: ultrasound — sonographic evaluation of intestinal blood flow

SUMMARY:
The purpose of the study is to determine whether packed red blood cell (PRBC) transfusion affects intestinal blood flow of premature infants during feedings and if so, whether return of normal intestinal blood flow pattern occurs within 48 hours of blood transfusion.

Abnormal intestinal responses to the feedings (insufficient postprandial blood flow increase in order to digest given feeding volume or overall decrease of intestinal blood flow) may predispose infants to feeding intolerance and to serious intestinal disease called necrotizing enterocolitis (NEC).

Patent ductus arteriosus (PDA) is a relatively common heart condition found in young preterm infants that can lead to decreased blood flow in different organs, including intestines. Thus, the determination of the presence or absence of PDA is an important part of the study, since it can be a relevant confounding variable.

In this study, the investigators will assess intestinal blood flow by using sonogram to measure velocity through the superior mesenteric artery (SMA), the artery supplying most of the intestine, both pre- and 45 minutes post feeding. The investigators will also use echocardiogram to determine the presence or absence of PDA. Each set of measurements will be done immediately before and after the transfusion, and again 24 and 48 hours after the transfusion.

Specific Hypothesis: The investigators hypothesize that infants will have attenuated postprandial blood flow velocities in immediate posttransfusion state when compared to the pretransfusion values. The investigators further hypothesize that normal, pretransfusion postprandial blood flow velocities will be achieved 48 hrs after the blood transfusion.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is the death of intestinal tissue. It most often affects premature or sick babies. NEC occurs when the lining of the intestinal wall dies and the tissue falls off. NEC is a known complication of prematurity with high morbidity and mortality. About 7 to 13% of all very low birth weight infants admitted to Neonatal Intensive Care Units (NICU) develop NEC, with mortality ranging from 10 to 44% (1,2,3).

NEC is considered a multifactorial disorder converging on a common final clinical presentation associated with several etiologic mechanisms, including ischemia (eg reperfusion), infection (eg, gut colonization), mechanical injury (eg, viscosity, embolic), iatrogenic factors (eg catheters, excessive enteral feeding), and immunological barrier dysfunction (1,13,4,5) To date, there is no single, unifying consensus on causation (6).

Newly, the association between NEC and Packed Red Blood Cell (PRBC)transfusion has been a subject of recent debate. Several retrospective studies report increased incidence of NEC 22 hrs (7) or 48-72 hrs after PRBC transfusion (8) and increased odds of NEC development within 48 hrs posttransfusion (9). Singh, measuring the strength of association between the NEC and PRBC transfusion describes the association as strong < 24hrs, less strong < 48 hrs and absent at 96 hrs (10). Importantly, the majority of the infants in these studies were stable premature neonates on full enteral feeds, who decompensated and developed NEC after being transfused.

Based on poor or no evidence, many NICUs are implementing policy not to feed premature infants during the blood transfusion (11). A small recent prospective trial (8) reported decreased incidence of NEC (from 5.3 to 1.3%) when feeds are withheld during the transfusion. Similarly, the limited investigation of the superior mesenteric artery (blood vessel that supplies the greatest volume of blood to the intestinal tract) blood flow velocities (SMA BFV) revealed that the expected post-prandial increase in SMA BFV disappeared following the PRBC, placing the fed neonates receiving blood transfusion at higher risk for NEC (12).

This initial study had several major limitations, such as enrolling larger and more mature preterm neonates at lesser risk for PRBC transfusion related NEC, excluding infants with patent ductus arteriosus (PDA), common clinical condition in preterm neonates, losing 11 out of 22 patients for follow up studies (hence "normalization" of post-prandial blood flow velocities and finding potentially safe time point for feeds reintroduction could not be suggested by the study results) and using relatively less commonly transfused PRBC volumes over longer period of time.

In this study, the investigators intend to further their understanding of the hemodynamic consequences of PRBC transfusion in very low birth weight (VLBW) neonates by evaluating pre-and post-prandial SMA BFV in neonates who are not fed during the transfusion at different time points and correlate those with relevant clinical outcome measures. The investigators anticipate that the results from this study will be used by clinicians to help guide them in making decisions regarding the safety of administering PRBC transfusion in VLBW neonates.

ELIGIBILITY:
Inclusion Criteria:

* birth weight ≤ 1500 gm
* singleton and multiple gestation
* small and appropriate birth weight for gestational age
* tolerance of ≥ 20 ml/kg/day of feeding volumes over 30 minutes or less
* at least 14 days of age and ≤ 35 6/7 weeks corrected gestational age at time of transfusion.
* Expected age range of 0-3 months is based on expected age of extremely low birth weight infants at limit (35 6/7 weeks) of corrected gestational age.

Only those infants who receive transfusion at < or equal to 35 weeks will undergo the PDA/SMA and BFV procedures and have data included in analysis.

Exclusion Criteria:

* major congenital or chromosomal anomalies
* presence of congenital heart disease (minus patent ductus arteriosus
* presence of shock
* presence of vasopressor use
* presence of severe lung disease
* concurrent treatment with antibiotics for sepsis
* history of NEC Bell stage 2 or greater
* Infants experiencing changes in vital signs or oxygen level drop needing intervention (such as oxygen increase or stimulation) will have studies discontinued and will be excluded from further analysis.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates (≤1500 grams of birth weight) of singleton and multiple births who are admitted to the NICU at Cardinal Glennon Children's Hospital and who are tolerating ≥ 20 ml/kg/day of feeding volume run over 30 minutes or less; both males and females of all ethnic groups.
  Very Low Birth Weight (VLBW) neonates will be studied since morbidities such as transfusion related acute gastrointestinal injury and/or necrotizing enterocolitis, PDA and feeding intolerance most frequently occur in this group.
  Because the need to ensure parental comprehension prior to consent documentation, parents who, in the judgement of the attending physician and/or research team members, do not have an adequate command of the English language will not be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Assessing intestinal blood flow by comparing superior mesenteric artery velocities in preterm neonates before and after packed red blood cell transfusion using sonogram. | Measurements are obtained both before and 45 minutes after feeding prior to transfusion; again before and after feeding after transfusion and again at 24 and 48 hours after the transfusion.
  Prospective investigation of pre- and post-prandial (45 minutes after feeding completion) SMA BVF in preterm neonates before and after blood transfusion. The pretransfusion SMA BFV measurements (pre- and post-prandial) are done during the last feeding before the transfusion; the postransfusion SMA BFV (pre- and post-prandial) measurements are done during the first feeding immediately following the blood transfusion and again during the feedings 24 and 48 hrs after the transfusion (Total of 8 SMA BFV assessments).

SECONDARY OUTCOMES:
To determine whether packed red blood cell transfusion affects patent ductus arteriosus status of the subjects using Echocardiogram to determine the presence or absence of PDA. | Each set of measurements will be done immediately before and after the transfusion, and again 24 and 48 hours after the transfusion.
  Before each SMA BFV measurement prior to feeding, the investigators will determine the presence or absence of PDA, since the presence of PDA can affect SMA BFV (total of 4 PDA studies for each enrolled subject).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Havranek, MD, Study Director — Saint Louis University, Cardinal Glennon Children's Hospital; Aaron Pitzele, MD, Principal Investigator — Saint Louis University, Cardinal Glennon Children's Medical Center
Locations (1):
- Cardinal Glennon Children's Hospital / Saint Louis University, St Louis, Missouri, United States

REFERENCES:
- [Background] Stoll BJ. Epidemiology of necrotizing enterocolitis. Clin Perinatol. 1994 Jun;21(2):205-18. doi: 10.1016/S0095-5108(18)30341-5. PMID 8070222
- [Background] Luig M, Lui K; NSW & ACT NICUS Group. Epidemiology of necrotizing enterocolitis--Part II: Risks and susceptibility of premature infants during the surfactant era: a regional study. J Paediatr Child Health. 2005 Apr;41(4):174-9. doi: 10.1111/j.1440-1754.2005.00583.x. PMID 15813870
- [Background] Holman RC, Stoll BJ, Clarke MJ, Glass RI. The epidemiology of necrotizing enterocolitis infant mortality in the United States. Am J Public Health. 1997 Dec;87(12):2026-31. doi: 10.2105/ajph.87.12.2026. PMID 9431297
- [Background] La Gamma EF, Browne LE. Feeding practices for infants weighing less than 1500 G at birth and the pathogenesis of necrotizing enterocolitis. Clin Perinatol. 1994 Jun;21(2):271-306. PMID 8070227
- [Background] Uauy RD, Fanaroff AA, Korones SB, Phillips EA, Phillips JB, Wright LL. Necrotizing enterocolitis in very low birth weight infants: biodemographic and clinical correlates. National Institute of Child Health and Human Development Neonatal Research Network. J Pediatr. 1991 Oct;119(4):630-8. doi: 10.1016/s0022-3476(05)82418-7. PMID 1919897
- [Background] Obladen M. Necrotizing enterocolitis--150 years of fruitless search for the cause. Neonatology. 2009;96(4):203-10. doi: 10.1159/000215590. Epub 2009 Apr 29. PMID 19407465
- [Background] Mally P, Golombek SG, Mishra R, Nigam S, Mohandas K, Depalhma H, LaGamma EF. Association of necrotizing enterocolitis with elective packed red blood cell transfusions in stable, growing, premature neonates. Am J Perinatol. 2006 Nov;23(8):451-8. doi: 10.1055/s-2006-951300. Epub 2006 Sep 28. PMID 17009195
- [Background] El-Dib M, Narang S, Lee E, Massaro AN, Aly H. Red blood cell transfusion, feeding and necrotizing enterocolitis in preterm infants. J Perinatol. 2011 Mar;31(3):183-7. doi: 10.1038/jp.2010.157. Epub 2011 Jan 20. PMID 21252964
- [Background] Paul DA, Mackley A, Novitsky A, Zhao Y, Brooks A, Locke RG. Increased odds of necrotizing enterocolitis after transfusion of red blood cells in premature infants. Pediatrics. 2011 Apr;127(4):635-41. doi: 10.1542/peds.2010-3178. Epub 2011 Mar 14. PMID 21402638
- [Background] Singh R, Visintainer PF, Frantz ID 3rd, Shah BL, Meyer KM, Favila SA, Thomas MS, Kent DM. Association of necrotizing enterocolitis with anemia and packed red blood cell transfusions in preterm infants. J Perinatol. 2011 Mar;31(3):176-82. doi: 10.1038/jp.2010.145. Epub 2011 Jan 27. PMID 21273983
- [Background] Agwu JC, Narchi H. In a preterm infant, does blood transfusion increase the risk of necrotizing enterocolitis? Arch Dis Child. 2005 Jan;90(1):102-3. doi: 10.1136/adc.2004.051532. No abstract available. PMID 15613530
- [Background] Krimmel GA, Baker R, Yanowitz TD. Blood transfusion alters the superior mesenteric artery blood flow velocity response to feeding in premature infants. Am J Perinatol. 2009 Feb;26(2):99-105. doi: 10.1055/s-0028-1090595. Epub 2008 Nov 19. PMID 19021097
- [Background] Simmonds A, LaGamma EF. Addressing the